CLINICAL TRIAL: NCT04554719
Title: Clinical Application of Fibroblast Activation Protein PET/MRI for Diagnosis and Staging
Brief Title: Clinical Application of Fibroblast Activation Protein PET/MRI for Diagnosis and Staging in Malignant Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0290
Record Dates: First submitted 2020-09-02; First posted 2020-09-18 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-02

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Gallium-68; Positron-Emission Tomography; Magnetic Resonance Spectroscopy; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTA-FAPI PET/MR (Experimental): Investigators select subjects from patients with suspected or diagnosed or treated malignant tumors who have completed 18F-FDG PET/CT imaging, focusing on malignant tumors with poor results of FDG PET/CT imaging, such as brain tumors, liver tumors, digestive system tumors and peritoneal, greater omentum, and mesenteric metastatic tumors. Patients undergo 68Ga-DOTA-FAPI PET/MR imaging within one week.
  Interventions: Drug: 68Ga-DOTA-FAPI; Device: PET/MR; Device: PET/CT

INTERVENTIONS:
Drug: 68Ga-DOTA-FAPI — Intravenous access is established in advance, intravenous bolus injection, 68Ga-DOTA-FAPI dose is about 1.85-3.7 MBq/kg body weight (0.05-0.1 mCi/kg), rinsed with 0.9% saline, and hydrated after drinking more water.
  Other Names: gallium-68 (68Ga)-Fibroblast activation protein inhibitor (FAPI)
Device: PET/MR — Each subject undergoes PET/MR imaging within 40-60 minutes after injection.
  Other Names: Positron Emission Tomography/Magnetic Resonance
Device: PET/CT — Each subject undergoes PET/CT imaging within 40-60 minutes after injection.
  Other Names: Positron Emission Tomography/Computed Tomography

SUMMARY:
Positron emission tomography (PET) molecular imaging provides a valuable tool for the diagnosis and differential diagnosis, staging of various tumors. Malignant tumor is composed of tumor cells and tumor stroma, which occupies the vast majority of the tumor. Cancer-associated fibroblasts (CAF) are an important part of the tumor stroma. Fibroblast activation protein (FAP) is over-expressed in CAF, which is closely related to tumor growth, invasion, metastasis, immunosuppression and prognosis; and the expression level of FAP in normal tissues and organs is very low. So it becomes an excellent target for cancer diagnosis and treatment. Radionuclide-labeled fibroblast activation protein inhibitors (FAPI) that specifically target to FAP as a tracer for PET imaging can be applied for targeted diagnosis and treatment of cancer. Recently, some studies have found that gallium-68 (68Ga) -FAPI as a new novel positron tracer has shown to be with good application potential. In this prospective study, the investigators will use integrated PET/MR, and PET/CT with the agent 68Ga-FAPI and conventional imaging agent [F-18] fluorodeoxyglucose (18F-FDG) to diagnose and stage various cancers, the aim is to make up for the deficiency in FDG PET imaging in the diagnosis and staging of some cancers.

DETAILED DESCRIPTION:
Positron emission tomography (PET) molecular imaging provides a valuable tool for the diagnosis and differential diagnosis, staging of various tumors. The most commonly used imaging agent is [F-18] fluorodeoxyglucose (18F-FDG), known as the "molecule of the century". However, in some low-grade gliomas, mucinous adenocarcinoma, bronchoalveolar carcinoma, primary hepatocellular carcinoma, renal clear cell carcinoma and some prostate cancers, factors such as the low expression level of tumor glucose transporter but high level of dephosphorylation, and the low number of tumor cells in tumor tissues can also be manifested as low absorption of 18F-FDG; in addition, 18F-FDG PET has limited ability to detect small lesions in some organs such as brain, liver, and kidneys that have physiological uptake or excretion of FDG with the relatively high background signal; moreover, the distribution of FDG in the body is easily affected by blood sugar. These factors limit the application value of 18F-FDG PET/CT in the differential diagnosis and staging of some malignant tumors.

A malignant tumor is composed of tumor cells and tumor stroma, which occupies the vast majority of the tumor. Cancer-associated fibroblasts (CAF) are an important part of the tumor stroma. Fibroblast activation protein (FAP) is over-expressed in CAF, which is closely related to tumor growth, invasion, metastasis, immunosuppression and prognosis; and the expression level of FAP in normal tissues and organs is very low, so it becomes an excellent target for cancer diagnosis and treatment. The use of radionuclide-labeled fibroblast activation protein inhibitors (FAPI) that specifically bind to FAP as a tracer for PET imaging can be applied for targeted diagnosis and treatment of cancer. Recently, some studies have found that gallium-68 (68Ga) -FAPI as a new novel positron tracer has shown to be with good application potential. The probe has very low background uptake in different types of cancer, so it can obtain high image contrast and clear tumor boundary. And it has good stability in serum and can be quickly removed from normal organs in vivo. In this project, we plan to apply the integrated PET / MR imaging of fibroblast activating protein (FAP) in the diagnosis and staging of malignant tumors, and compare it with 18F-FDG PET / CT imaging, so as to make up for the deficiency in FDG PET imaging in the diagnosis and staging of some tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or diagnosed or treated malignant tumors who have completed 18F-FDG PET/CT imaging.
* Subjects are able to understand and sign the informed consent voluntarily, with good compliance.

Exclusion Criteria:

* Acute systemic diseases and electrolyte disorders.
* Pregnant or lactating women.
* Patients refuse to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 68Ga-DOTA-FAPI PET/MR for diagnosis and staging in some malignant tumors. | 2 years
  For subjects with suspected or diagnosed or treated malignant tumors who have completed 18F-FDG PET/CT imaging, diagnosis and staging results of 68Ga-DOTA-FAPI PET/MR, PET/CT will be compared to 18F-FDG PET/CT imaging, pathology, clinical and follow-up result.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin C, Song Y, Gai Y, Ruan W, Liu Q, Liu F, Zheng D, Zhang P, Liu H, Zhang T, Tao K, Lan X. Gallium-68-labeled fibroblast activation protein inhibitor PET in gastrointestinal cancer: insights into diagnosis and management. Eur J Nucl Med Mol Imaging. 2022 Oct;49(12):4228-4240. doi: 10.1007/s00259-022-05847-0. Epub 2022 Jun 3. PMID 35657428
- [Derived] Qin C, Song Y, Liu X, Gai Y, Liu Q, Ruan W, Liu F, Hu F, Lan X. Increased uptake of 68Ga-DOTA-FAPI-04 in bones and joints: metastases and beyond. Eur J Nucl Med Mol Imaging. 2022 Jan;49(2):709-720. doi: 10.1007/s00259-021-05472-3. Epub 2021 Jul 9. PMID 34241652
- [Derived] Qin C, Liu F, Huang J, Ruan W, Liu Q, Gai Y, Hu F, Jiang D, Hu Y, Yang K, Lan X. A head-to-head comparison of 68Ga-DOTA-FAPI-04 and 18F-FDG PET/MR in patients with nasopharyngeal carcinoma: a prospective study. Eur J Nucl Med Mol Imaging. 2021 Sep;48(10):3228-3237. doi: 10.1007/s00259-021-05255-w. Epub 2021 Feb 20. PMID 33609152
- [Derived] Zhang X, Song W, Qin C, Liu F, Lan X. Non-malignant findings of focal 68Ga-FAPI-04 uptake in pancreas. Eur J Nucl Med Mol Imaging. 2021 Jul;48(8):2635-2641. doi: 10.1007/s00259-021-05194-6. Epub 2021 Jan 15. PMID 33452634